CLINICAL TRIAL: NCT01749332
Title: A Pilot Study of Perihepatic Phlebotomy During Hepatic Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-236
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Liver Cancer
Keywords: blood draw; Perihepatic Phlebotomy; 12-236
MeSH Terms: conditions — Liver Neoplasms

ARMS (1):
- Pts having liver or colon surgery (Experimental): Blood will be obtained from patients at the time of laparotomy for hepatic resection and/or hepatic arterial infusion pump placement, or pancreatic head resection . Blood will be drawn from a peripheral vein or artery (when an arterial catheter is present), the portal vein, and suprahepatic IVC and given to a research assistant and placed on ice followed by immediate processing. Total amount of blood drawn will not exceed fifty milliliters (50ml).
  Interventions: Other: Perihepatic Phlebotomy

INTERVENTIONS:
Other: Perihepatic Phlebotomy

SUMMARY:
The purpose of this study is to draw blood from vessels near the liver in patients undergoing liver surgery. This will be performed in both patients with cancer in order to learn more about circulating tumor cells, proteins and DNA mutations in the blood.

The blood in patients with colorectal cancer with liver metastases will be compared to blood taken from patients that do not have cancer that do not have cancer.

Inclusion of patients with benign pathology will allow for the establishment of "normal" values which currently do not exist. We will then study whether tumor mutations can be used to predict recurrence and survival patterns.

ELIGIBILITY:
Inclusion Criteria:

* All patients with resectable CRLM without extrahepatic metastases confirmed by tissue diagnosis or radiologic exam who are undergoing hepatic resection.
* All patients undergoing hepatic arterial infusion pump placement with or without without hepatic resection.
* Patients may have synchronous or metachronous CRLM
* Patients may have received prior cytotoxic (must be off for at least 2 weeks prior to surgery) or anti-angiogenic therapy (must be off for at least 6 weeks prior to surgery). Specific drugs are listed below.
* 5-FU based chemotherapy - 2 weeks off
* Bevacizumab - 6 weeks off
* Cetuximab or panitumumab - 2 weeks off
* Control patients will include patients consented for pancreaticoduodenectomy for benign or pre-neoplastic lesions. If lesions assumed to be benign turn out to be malignant on final pathology, the blood will be discarded and the patient replaced.
* Patients undergoing a two-stage hepatectomy resection, or who are reevaluated for a second hepatectomy, will be considered for reenrollment to protocol

Exclusion Criteria:

* Evidence of extra-hepatic disease on pre-operative imaging or at operative exploration, excluding the primary colorectal tumor
* Those with known bleeding or clotting diatheses
* Patients diagnosed with chronic inflammatory diseases such as lupus, rheumatoid arthritis, psoriasis, ulcerative colitis, Crohns disease, etc.
* Pre- or intra-operative evidence of portal vein thrombosis or hypertension
* Patients who have taken immune modulating agents in the past 8 weeks including steroids, anti-TNF-α, interferon etc. Patients taking a single dose of Decadron as part of a chemotherapy regimen will not be excluded from the study.
* Patients who take daily anti-inflammatory medications such as COX-2 inhibitors or high dose NSAIDs. Patients taking a daily aspirin or acetaminophen or occasional anti-inflammatory medications will not be excluded from the study.
* If at the discretion of the operating surgeon, blood acquisition would lead to undue morbidity, the patient will be excluded and replaced
* Attending physicians authorized to obtain informed consent may exercise discretion in excluding individuals for appropriate medical or other reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
ctDNA differences | once at the time of surgery
  to collect preliminary data on perihepatic and peripheral ctDNA differences between prehepatic and posthepatic sites in patients with and without primary colorectal cancers in place.

SECONDARY OUTCOMES:
collect preliminary data | 1 year
  to correlate perihepatic and peripheral ctDNA mutation with recurrence and survival patterns. This will be performed by log-ranks tests of recurrence free survival and overall survival for each gene and possibly for the most common combinations of mutations

CONTACTS AND LOCATIONS:
Overall Officials: Michael D'Angelica, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/